CLINICAL TRIAL: NCT06464614
Title: A Double-arm, Non-randomized Controlled, Open-label Clinical Study of Adebrelimab in Combination With Apatinib and Chemotherapy/Chemoradiotherapy in Immuno-experienced Second-line Esophageal Squamous Cell Carcinoma.
Brief Title: Adebrelimab in Combination With Apatinib and Chemotherapy/Chemoradiotherapy in Immuno-experienced Second-line ESCC.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADE-ESCC-02
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — apatinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adebrelimab＋Apatinib＋Radiotherapy＋Investigator chosen chemotherapy (ICC) (Experimental): Adebrelimab（1200mg，d1 q3w, continuous medication until disease progression, intolerable toxicity, or withdrawal due to other reasons），Apatinib (250mg，d1-21，q3w), Radiotherapy， Investigator chosen chemotherapy (ICC)
  Interventions: Drug: Adebrelimab; Drug: Apatinib; Drug: Investigator chosen chemotherapy (ICC); Radiation: Radiotherapy
- Adebrelimab＋Apatinib＋Investigator chosen chemotherapy (ICC) (Experimental): Adebrelimab（1200mg，d1 q3w, continuous medication until disease progression, intolerable toxicity, or withdrawal due to other reasons），Apatinib (250mg，d1-21，q3w), Investigator chosen chemotherapy (ICC)
  Interventions: Drug: Adebrelimab; Drug: Apatinib; Drug: Investigator chosen chemotherapy (ICC)

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab 1200mg，d1，q3w, until disease progression or unacceptable toxicity
  Other Names: SHR-1316
Drug: Apatinib — Apatinib 250mg，d1-21，q3w, until disease progression or unacceptable toxicity
  Other Names: Apatinib capsule
Drug: Investigator chosen chemotherapy (ICC) — Nab-paclitaxel: 125mg/m2 intravenously, D1, D8, q3w, 4-6 cycles;Intravenous infusion of 100 mg, D1, qw is used at the same time as radiotherapy.
  Ilinotecan: 125mg/m2 intravenously, D1, D8, q3w, 4-6 cycles; Capecitabine, 625 mg/m2 orally, d1-14, q3w; continued until disease progression, intolerable toxicity, or withdrawal due to other reasons; when synchronized with radiotherapy, 625mg/m2, bid, oral, d1-5, qw.
  Other Names: Albumin-paclitaxel
Radiation: Radiotherapy — Radiotherapy mode: IMRT for the primary lesion and SBRT for the metastasis; If the patient has symptoms of dysphagia, the radiation dose is 1.8 Gy×28 F or 2 Gy×25 F, d1-5 5 times a week; If oligometastatic lesions occur in the body: the radiation dose is 8 Gy×5F, d1-5; If oligometastatic lesions occur in the brain, the radiation dose is 7 Gy×5F, d1-5.
  Arms: Adebrelimab＋Apatinib＋Radiotherapy＋Investigator chosen chemotherapy (ICC)

SUMMARY:
To assess the efficacy and safety of adebrelimab in combination with apatinib mesylate and chemoradiotherapy in immuno-experienced second-line esophageal squamous cell carcinoma (with symptomatic dysphagia or oligometastatic disease)，and to evaluate the efficacy and safety of adebrelimab in combination with apatinib mesylate and chemoradiotherapy in immuno-experienced second-line esophageal squamous cell carcinoma (without symptomatic dysphagia or oligometastatic disease).

DETAILED DESCRIPTION:
The treatment of advanced second-line esophageal squamous cell carcinoma has always been mainly chemotherapy. Since 2019, a number of phase III clinical trials (ESCORT, KEYNOTE-181, RATIONALE 302, ATRACTION-3, etc.) have confirmed that there is a significant difference in OS between the immune monotherapy group and the chemotherapy group, and immunotherapy can bring better survival benefits. Although the above studies have brought new possibilities for second-line patients with advanced esophageal cancer, the results of the study show that the response rate of immune monotherapy is limited, with a single-agent ORR of about 13%-20%, mPFS of about 2 months, and mOS about 8 months. Therefore, finding a suitable combination therapy model to further improve the efficacy of advanced second-line esophageal cancer has gradually become a research hotspot in recent years. In recent years, many experts have also made a lot of explorations. The combination of anti-angiogenic drugs and immunotherapy drugs can be synergistic.

Dysphagia is a major symptom in patients with esophageal cancer, leading to significant nutritional deficiencies, pain, and subsequent deterioration in quality of life. Management of dysphagia is a key goal of esophageal cancer treatment, along with the need to improve nutritional status and quality of life, which may have a positive impact on the overall prognosis of patients. Current treatment methods for dysphagia include esophageal dilation, endoluminal stenting, systemic chemotherapy, external beam radiotherapy (EBRT), brachytherapy, and concurrent chemoradiotherapy (CTRT). At present, there is no consensus on how to better manage this symptom with these treatment regimens, and more research is needed to continue to explore.

To assess the efficacy and safety of adebrelimab in combination with apatinib mesylate and chemoradiotherapy in immuno-experienced second-line esophageal squamous cell carcinoma (with symptomatic dysphagia or oligometastatic disease), and to evaluate the efficacy and safety of adebrelimab in combination with apatinib mesylate and chemoradiotherapy in immuno-experienced second-line esophageal squamous cell carcinoma (without symptomatic dysphagia or oligometastatic disease).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years old, male or female; 2. Esophageal squamous cell carcinoma confirmed by histology or cytology; 3. Patients who have progressed or are intolerant to first-line chemotherapy combined with immunotherapy (chemotherapy regimen can include platinum, purple shirt or fluorouracil as the basis, etc.) (progression of maintenance therapy after first-line chemotherapy combined with immunization can also be included).

  4. Cohort A: Subjects who have at least one of the following two conditions will be treated with adebelimab combined with apatinib mesylate and chemoradiotherapy;
  1. Symptomatic dysphagia, Mellow score ≥1 (Mellow score: 0 = able to eat all solid foods, 1 = only partially solid foods, 2 = able to eat soft foods, 3 = only able to drink liquids, 4 = complete dysphagia);
  2. Hypometastatic disease: Oligometastatic disease is considered when there are ≤ 3 metastases in the liver, lungs, retroperitoneal lymph nodes, adrenal glands, soft tissues, bones, or brain. In addition, after receiving a median of 18 weeks of systemic therapy, metastatic lesions are considered to be oligometastatic lesions at the time of restaging if they do not progress or only progress in size. If the number of lesions increases when restaged after systemic therapy, it is not considered oligometastatic disease.

     Cohort B: If the subjects do not have the above conditions, they will be treated with adebelimab in combination with apatinib mesylate and chemotherapy; 5. Have at least one measurable lesion according to the Efficacy Evaluation Criteria in Solid Tumors (RECIST 1.1); 6.ECOG：0～1； 7. Expected survival≥12 weeks; 8. The blood routine and biochemical indexes of the subjects within 7 days before enrollment meet the following criteria:

     a. Hemoglobin ≥90g/L, absolute neutrophil count (ANC) ≥ 1.5×109/L, platelet ≥ 100×109/L (patients must not have received blood transfusion or growth factor support within 14 days of blood sample collection); b. ALT, AST ≤ 2.5 times the upper limit of normal (ULN); ALP ≤ 2.5 times ULN; c. Serum total bilirubin < 1.5 times ULN (patients with Gilbert syndrome can be enrolled if total bilirubin < 3 times ULN); d. Serum creatinine < 1.5 times ULN or estimated glomerular filtration rate ≥60ml/min/1.73m2; e. Serum albumin≥30g/L; International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN, unless the patient is receiving anticoagulant therapy and the PT value is within the range of anticoagulant intended treatment; Activated partial thromboplastin time (APTT) ≤ 1.5 times ULN. 9. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ low limit of normal (50%).

  10. Females of childbearing potential should agree to use contraception (such as intrauterine device, contraceptive pills or condoms) during the study and for 6 months after the end of the study, have a negative serum or urine pregnancy test within 7 days prior to study enrollment and must be non-lactating patients, and males should agree to use contraception during the study and for 6 months after the end of the study period; 11. No serious concomitant disease that makes the survival time < 5 years; 12. Subjects voluntarily joined this study, signed the informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* 1. Patients have any active autoimmune disease or history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; patients with vitiligo; asthma that has been completely relieved in childhood and does not require any intervention in adulthood can be included; asthma patients requiring medical intervention with bronchodilators cannot be included); 2. The patient is using immunosuppressants, or systemic hormone therapy to achieve the goal of immunosuppression (dose> 10mg/day prednisone or other effective hormones), and continues to use it within 2 weeks before enrollment; 3. Patients with esophageal squamous cell carcinoma whose primary lesion is active hemorrhage; 4. Those with a variety of factors that affect oral medication (such as inability to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.); 5. Patients with brain metastases with symptoms or symptomatic control time of less than 3 months; 6. Patients with any severe/uncontrolled disease, including: patients with unsatisfactory blood pressure control (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100 mmHg); Patients with grade I or grade myocardial ischemia or myocardial infarction, arrhythmias (including QT interval ≥480ms) and grade I cardiac insufficiency, active or uncontrolled serious infections, liver disease such as decompensated liver disease, active hepatitis B (HBV-DNA≥ 104 copies/ml or 2000IU/ ml) or hepatitis C (positive for hepatitis C antibody and HCV-RNA above the lower limit of detection of the analytical method), urinalysis shows urine protein ≥++, and 24-hour urine protein quantification >1.0g; 7. Long-term unhealed wounds or fractures; 8. Pulmonary hemorrhage with NCI CTCAE grade >1 within 4 weeks prior to enrollment; bleeding from other sites with NCI CTCAE grade >2 within 4 weeks prior to enrollment; patients with bleeding tendencies (such as active peptic ulcers) or patients who are receiving thrombolytic or anticoagulant therapy such as warfarin, heparin, or their analogues; 9. Patients who have had arterior/venous thrombotic events within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism; 10. Patients whose imaging shows that the tumor has invaded important blood vessels or who are judged by the investigator to have a high probability of invading important blood vessels during the follow-up study period, causing fatal hemorrhage; 11. Pregnant or lactating women; 12. Patients with other malignant tumors within 5 years (except for basal cell carcinoma of the skin and carcinoma in situ of the cervix that have been cured); 13. Patients with a history of psychotropic drug abuse who cannot be abstained from or patients with mental disorders; 14. Patients who have participated in clinical trials of other drugs within four weeks; 15. According to the judgment of the investigator, patients with concomitant diseases that seriously endanger the safety of patients or affect the completion of the study; 16. Those who, in the opinion of the investigator, are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival，PFS | 9 months
  Time from randomization to patient's tumor progression or death

SECONDARY OUTCOMES:
Objective Response Rate，ORR | 1 year
  The proportion of patients whose tumor shrinks to a certain amount and remains for a certain period of time
Overall survival,OS | 1 year
  The time from the beginning of randomization to death due to any cause.
Duration of Response,DoR | 1 year
  The time from the first assessment of the tumor as CR or PR to the first assessment of PD (Progressive Disease) or death from any cause.
Disease control rate,DCR | 1 year
  The proportion of patients whose tumors have shrunk or stabilized and remain for a certain period of time (mainly for solid tumors), including cases of complete response (CR), partial response (PR) and stable disease (SD).
Time to response | 1 year
  Time from randomization to the achievement of the first objective response
1-year OS rate | 1 year
  Percentage of patients who are still alive after 1 year
9-month survival rate | 1 year
  Percentage of patients who are still alive after 9-month

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China